CLINICAL TRIAL: NCT02011763
Title: Safety of Two Doses of Avaxim® 80U Pediatric (Inactivated Hepatitis A Vaccine) Administered 6 Months Apart in Healthy Toddlers, Children and Adolescents Aged 12 Months to 15 Years in China
Brief Title: Safety of Two Doses of Avaxim® 80U Pediatric (Inactivated Hepatitis A Vaccine) in Toddlers, Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HAF87; U1111-1127-7652 (Other: WHO)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis A; Hepatitis A Virus
Keywords: Hepatitis A; hepatitis A virus; Avaxim® 80U Pediatric
MeSH Terms: conditions — Hepatitis A; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Toddlers, children and adolescents aged 12 months to 15 years
  Interventions: Biological: Avaxim 80U Pediatric: Inactivated Hepatitis A Virus

INTERVENTIONS:
Biological: Avaxim 80U Pediatric: Inactivated Hepatitis A Virus — 0.5 mL, Intramuscular (2 injection 6 months apart)
  Other Names: Avaxim 80U Pediatric

SUMMARY:
The aim of this study is to describe the safety profile of Avaxim 80U Pediatric, in order to confirm the good safety profile of the vaccine.

Primary objective:

* To describe the safety of Avaxim 80U Pediatric after each dose of vaccine administered 6 months apart, in subjects aged 12 months to 15 years.

DETAILED DESCRIPTION:
Eligible participants aged 12 months to 15 years and 5 months (185 months) at enrollment will receive two doses of vaccine for the prevention of hepatitis A (6 months apart), and will be followed up for safety until 30 days after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 185 months (approximately 15 years and 5 months) on the day of inclusion
* Informed consent form has been signed and dated by the subject aged 12 years old and above (based on local regulations), and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative
* Subject and parent / legally acceptable representative are able to attend all schedule visits and to comply with all trial procedures
* Subjects aged less than 2 years only: Born at full term of pregnancy (≥ 37 weeks) and/or with a birth weight ≥ 2.5 kg.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks preceding or following any trial vaccination
* Previous vaccination against Hepatitis A with either the trial vaccine or another Hepatitis A vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of Hepatitis A infection, confirmed either clinically, serologically, or microbiologically
* At high risk for hepatitis A infection during the trial
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness / infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 355 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited injection site and systemic events and unsolicited adverse events following vaccination with Avaxim® 80U Pediatric (Inactivated Hepatitis A vaccine). | Day 0 up to Day 30 post vaccination
  Participants aged ≤ 23 months, Solicited injection site reactions: Tenderness, Redness, and Swelling; Solicited systemic reactions: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite, and Irritability. Participants 2 to 15 Years of Age: Solicited injection site reactions: Pain, Redness, and Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia. Unsolicited adverse events, including serious adverse events will also be collected for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Beijing, China

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com